CLINICAL TRIAL: NCT04759066
Title: Assessment of an Alternative to Physical Wrist Restraints in Adult Intubated Patients in the Intensive Care Unit: The HEALiX™ Intubated Patient (IP) Pilot Study
Brief Title: The HEALiX™ Intubated Patient (IP) Pilot Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Primary investigator moved to a new institution.
Sponsor: Lancaster General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: HEALiX IP Pilot
Record Dates: First submitted 2021-02-12; First posted 2021-02-18 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Device Ineffective; Safety Issues
Keywords: self-extubation; non-restraint device; removal of lines

STUDY DESIGN:
Intervention Model Description: Single group descriptive pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Participants will wear HEALiX device
  Interventions: Device: HEALiX

INTERVENTIONS:
Device: HEALiX — HEALiX is a non-restraint patient safety device

SUMMARY:
The current standard of care for limiting the movement of mechanically ventilated critical care patients is the use of physical wrist restraints, which are both ineffective in preventing removal of invasive and adjunct respiratory support devices and have a multitude of negative physical and psychological consequences for the patient. The objective of the proposed research is to test an innovative device designed to allow more freedom of movement of mechanically ventilated patients without bending of the arms, thereby preventing removal of adjunct mechanical ventilation devices and invasive monitoring equipment.

ELIGIBILITY:
Inclusion Criteria:

* speak English
* legally authorized representative must speak English
* admitted by one of the services presiding over the selected intensive care units
* mechanically ventilated receiving analgesic-sedating medications
* have soft wrist restraints applied as part of their care plan documented in the medical record to reduce the risk of unplanned removal of medical devices

Exclusion Criteria:

* pregnant women
* prisoners
* patients who are in a medically induced coma or in a comatose state (Glasgow Coma Scale <8) for any reason

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Unplanned removal of devices | up to 2 weeks
  Frequency of unplanned removal of lines and self-extubation

SECONDARY OUTCOMES:
Ease of device use | up to 2 weeks
  Staff perception of ease of locating the correct size of the device, applying it, caring for the patient using HEALiX, cleaning it after use, and returning it for storage.
Availability of device | up to 2 weeks
  Number of times during the study period that the correct size of HEALiX is not available.
Alternate device use | up to 2 weeks
  Number of patients who have HEALiX device removed by staff and replaced by soft wrist restraints or other limb limiting application, and the reason for removal.
Ease of application | up to 1 week
  Proportion of incorrectly to correctly sized HEALiX applications
Acceptability of device | up to 1 week
  Average length of time for a member of the research team to discuss the HEALiX Pilot Study with a patient's family member in person and phone until decision is made about participation
Education around device | up to 12 weeks
  Length of time it takes to train the staff in the three participating Intensive Care Units

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Caplan, DNP-C, Principal Investigator — Penn Medicine Lancaster General Health
Locations (1):
- Lancaster General Health, Lancaster, Pennsylvania, United States